CLINICAL TRIAL: NCT02360761
Title: Surgical Treatment of Elderly Patients With Early Stage Non-small Cell Lung Cancer (STEPS): Comparison Between Sublobar Resection and Lobectomy - an Open, Multicenter, Randomized Phase III Clinical Trial
Brief Title: Surgical Treatment of Elderly Patients With cT1N0M0 Non-small Cell Lung Cancer Comparison Between Sublobar Resection and Lobectomy
Acronym: STEPS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Principal Investigator, Clinical Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1504
Record Dates: First submitted 2015-01-24; First posted 2015-02-11 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer;Elderly;Sublobar resection;Lobectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted; Thoracoscopy; Thoracotomy; Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lobectomy (Active Comparator): Patients undergo lobectomy by thoracotomy or thoracoscopy/Video assisted thoracoscopic surgery(VATS).
  Interventions: Procedure: VATS; Procedure: Thoracotomy
- Sublobar resection (Experimental): Patients undergo sublobar resection(wedge resection or anatomic segmentectomy) by thoracotomy or thoracoscopy/VATS.
  Interventions: Procedure: VATS; Procedure: Thoracotomy

INTERVENTIONS:
Procedure: VATS — Patients undergo lobectomy,wedge resection, or anatomical segmentectomy by thoracoscopic surgery or video assisted thoracoscopic surgery.
  Other Names: Thoracoscopy
Procedure: Thoracotomy — Patients undergo lobectomy, wedge resection, or anatomic segmentectomy by thoracotomy.
  Other Names: Open surgery

SUMMARY:
The role of sublobar resection(Wedge resection or anatomic segmentectomy) for small(≤ 2cm) early stage non-small cell lung cancer has been studied by Lung Cancer Study Group and is being studied by several ongoing trials. However, elderly patients(aged ≥70 years) in these trials is under-represented, as in most of the ongoing clinical trials. This study focuses on the elderly population of early stage lung cancer, and aims to investigate the outcome of lobectomy versus sublobar resection for peripheral stage I non-small cell lung cancer (NSCLC) in elderly patients.

DETAILED DESCRIPTION:
This randomized trial is to the best of our knowledge the first one designed to compare sublobar resection and lobectomy for elderly patients, in order to address these open questions:In patients aged 70 years or older and with clinical stage T1N0M0 NSCLC, (1) whether sublobar resection can achieve similar disease-free survival compared to lobectomy, (2) whether sublobar resection can reduce the postoperative mortality and morbidity,(3) whether sublobar resection can reserve better pulmonary function and quality of life for elderly patients of NSCLC?

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Preoperative criteria (contrast-enhanced Computed tomography scan)

  * Suspected non-small cell lung cancer
  * Clinical stage ⅠA, i.e. T1N0M0 (tumor diameter ≤3 cm, surrounded by visceral pleura, short-axis of lymph node <1 cm or cold lymph nodes on PET scan)
  * The maximum diameter of consolidation of the maximum tumor diameter (consolidation/tumor ratio, C/T ratio) is no less than 0.5 in sub-solid lesions
  * Eligible for sublobar resection with sufficient margin
* Intraoperative criteria

  * Histologically confirmed invasive NSCLC, i.e. NSCLC other than pre-invasive adenocarcinomas defined by The International Association for the Study of Lung Cancer (adenocarcinoma in situ, and minimally invasive adenocarcinoma)
  * Pathological exclusion of suspected lymph nodes involvement
  * Feasible to perform sublobar resection in terms of surgical margin requirement
* General criteria

  * Must sign informed consent by the patient or his/her entrusted party
  * Must complete 4-year mortality index and comprehensive geriatric assessment(CGA) if necessary
  * The physiological reservation can tolerate lobectomy

Exclusion Criteria:

* Unable to comply with the study procedure
* Past thoracic surgery history, except for diagnostic thoracoscopy
* Malignant tumor history within the past 5 years, except for the following conditions: cured skin basal cell carcinoma, superficial bladder carcinoma, and uterine cervix cancer in situ
* Any active systemic diseases including uncontrolled hypertension, unstable angina pectoris, newly onset of angina pectoris within recent 3 months, congestive heart failure (class II or plus of New York Heart Association, NYHA), myocardial infarction within recent 6 months, severe disease in the need of medication such as arrhythmia, liver, renal or metabolic diseases
* Uncontrollable infections
* Coexisting small cell lung cancer
* Psychiatric diseases diagnosed
* Other circumstances which is deemed inappropriate for enrollment by the researchers

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Time To Disease free survival Event | 3 years
  The time interval from randomization to the earliest onset of any of the following events: tumor recurrence, metastasis, or death caused by any reason.

SECONDARY OUTCOMES:
Percentage of Participants with Perioperative Complication and Death as a Measure of Safety. | 1 months
  Perioperative complication is defined as the complication occurred after surgery and before discharge, or within 30 days postoperatively. Death cases during this period should be recorded as perioperative death.
Hospitalization time after surgery in Participants | 1 months
  Defined as the time interval from the day of operation to discharge.
Intubation time after surgery in Participants | 1 months
  Defined as the time interval from the day of operation to extubation.
Time To Overall survival Event | 3 years
  The time interval from randomization to death from any cause.
Percentage of Participants With Local Recurrence and Metastasis Event | 3 years
  The ratio of local recurrence and metastasis in 3 years from the day of randomization
Postoperative pulmonary function | 3 years
  The Forced expiratory volume in one second and the forced vital capacity at 6-, 12- and 36-month post of the day of randomization.
Percentage of Participants With VATS procedure | 1 month
  The ratio of video assisted thoracoscopic surgery in each group.
Scores on the quality of life questionaires | 3 years
  The scores of the 6-, 12- and 36-month questionaire on quality of life post of the day of randomization.

OTHER OUTCOMES:
The scores of CGA and 4-year mortality index as a measure of predictive factor for the outcome of the elderly. | 3 years
  The scores of prospective CGA and 4-yr mortality index to predict the outcome of the elderly.
The total cost as a measure of the cost/benefit analysis | 3 years
  The cost/benefit analysis of sublobar resection versus lobectomy
The rate of pathologically noninvasive lung cancer with the radiologic character of C/T>0.5 | 1 month
  The radiologic character of C/T>0.5 has been considered as a pathologically noninvasive lung cancer. and the rate of pathologically noninvasive lung cancer will be used as a measure for the relation between the radiologic / pathologic character of primary non-small-cell lung cancer and prognosis.
The morbidity rate as a measure between the two different interventions as a Measure of Safety and Tolerability. | 3 years
  The morbidity rate after surgery for participants who underwent video-assisted thoracoscopic or open procedures a Measure of Safety and Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.M., Principal Investigator — Peking University People's Hospital
Locations (6):
- China (6):
  - Beijing Haidian Hospital, Beijing
  - Peking university people's hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sir Run Run Shaw Hospital, Hangzhao
  - The Affiliated Hospital of Qingdao University, Qingdao
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Derived] Yang F, Sui X, Chen X, Zhang L, Wang X, Wang S, Wang J. Sublobar resection versus lobectomy in Surgical Treatment of Elderly Patients with early-stage non-small cell lung cancer (STEPS): study protocol for a randomized controlled trial. Trials. 2016 Apr 7;17:191. doi: 10.1186/s13063-016-1312-6. PMID 27053091